CLINICAL TRIAL: NCT02387034
Title: The Effect on Swedish Physical Activity on Prescription (PAP) in Patients in Primary Care With Osteoarthritis in Knee or Hip - a RCT-study.
Brief Title: Swedish PAP in Osteoarthritis - a RCT Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Region Gävleborg (Other)
Responsible Party: Principal Investigator, Margareta Emtner, Assoiciate Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAVLE-2014-FAR
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Sedentary
Keywords: Osteoarthritis; Sedentary; Physical activity; Health related quality of life
MeSH Terms: conditions — Osteoarthritis; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity on prescription (PAP) (Experimental): Participants meet a physiotherapist for 60 minutes, get information about osteoarthritis, physical activity and weight control and a patient-centered counselling about physical activity related to the disease. It leads to a Swedish Physical activity on prescription (PAP). It is an individualized written prescription on physical activity and includes specific mode of physical activity. The patient is contacted by telephone or visit the physiotherapist after three weeks, three months and six months.
  Interventions: Behavioral: Physical activity on prescription
- General advice (Other): Participants meet a physiotherapist for 60 minutes, get information about osteoarthritis, physical activity and weight control and receive an intervention with general advice about being active with cardiovascular exercise such as walking, cycling or otherwise in 30 minutes three times a week and do strength training functional during the day such as walk in stairs and getting up from a chair without hand support.
  Interventions: Other: General advice

INTERVENTIONS:
Behavioral: Physical activity on prescription — Participants meet a physiotherapist for 60 minutes, get information about osteoarthritis, physical activity and weight control and a patient-centered counselling about physical activity related to the disease. It leads to a Swedish Physical activity on prescription (PAP). It is an individualized written prescription on physical activity and includes specific mode of physical activity. The patient is contacted by telephone or visit the physiotherapist after three weeks, three months and six months.
  Arms: Physical activity on prescription (PAP)
Other: General advice — Participants meet a physiotherapist for 60 minutes, get information about osteoarthritis, physical activity and weight control and receive an intervention with general advice about physical activity
  Arms: General advice

SUMMARY:
The purpose of this study is to determine whether an intervention with Physical activity on prescription (PAP) to individuals in primary care with knee or hip osteoarthritis would result in effects on physical activity level, physical capacity and quality on life.

The hypothesis is that patients with osteoarthritis in hip or knee will increase their level of physical activity significantly more with a PAP intervention compared to patients who only get general advice about physical activity.

DETAILED DESCRIPTION:
According to guidelines the recommended first-line management for people with osteoarthritis consist of exercise, information about osteoarthritis and if necessary, weight reduction. It is well documented that exercise has a positive effect on pain and physical function in these patients. Therefore, it is important to have methods to increase physical activity levels in these patients. It is not explored whether an intervention with PAP may lead to increased physical activity in patients with knee or hip osteoarthritis. The study will be a prospective, randomized, single-blind intervention study including 140 patients (70 patients/group). Patients will in a parallel design be randomized to intervention or control group. Both groups receive oral and written information about osteoarthritis and if necessary, advice on weight loss. The intervention group receives Swedish Physical activity on prescription. It is a patient-centered counselling about physical activity related to the disease. The counselling results in an individualized written prescription on physical activity including specific modes on physical activity. After three weeks, three months and six months they are offered a follow up which could be by telephone or personal meeting. During the follow up they discuss who the physical activity works out and plan new goals. The control group will receive an intervention with general advice about being active three times a week and do strength training functional during the day. Patients in the control group see the physiotherapist once.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically verified osteoarthritis in knee or hip
2. Sedentary (physical activity level, less than 150 minutes of moderate-intensity or less than 75 minutes of vigorous-intensity a week) includes

Exclusion Criteria:

1. Severe pain in hip or knee when walking
2. Other serious disorders causing problems when walking
3. Back injury causing pain in the leg
4. Cruciate ligament injury in the knee which causes severe dysfunction
5. Severe menisci injury
6. Total joint replacement in hip or knee
7. Unable to understand Swedish and follow verbal visual instructions

Study population: Patients who contact primary care center because of their hip or knee osteoarthritis and which is referred to the physical therapist. Seven health centers in Gävle include patients.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-06; Primary Completion 2017-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | Change from baseline to 6, 12, 24 months
  Physical activity will be measured with an activity monitor (accelerometer).

SECONDARY OUTCOMES:
Body composition | Change from baseline to 6,12, 24 months
  This will be measured with bio-impedance
Health related quality of Life , general | Change from baseline to 6,12,24 months
  This will be measured with EQ-5D
Health related quality of Life, disease specific | Change from baseline to 6,12,24 months
  HOOS, KOOS
Walking distance | Change from baseline to 6,12,24 months
  This will be measured with six-minute walk test
Leg muscle strength and function | Change from baseline to 6,12,24 months
  This will be measured with a standadised maximal step-up height test
Physical activity level | Change from baseline to 6,12,24 months
  Physical activity will be assessed by a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Karlsson, head, Principal Investigator — Primary health care in Gävle
Locations (1):
- Uppsala University, Uppsala, Sweden

REFERENCES:
- [Derived] Bendrik R, Kallings LV, Broms K, Kunanusornchai W, Emtner M. Physical activity on prescription in patients with hip or knee osteoarthritis: A randomized controlled trial. Clin Rehabil. 2021 Oct;35(10):1465-1477. doi: 10.1177/02692155211008807. Epub 2021 Apr 11. PMID 33843297